CLINICAL TRIAL: NCT04894448
Title: Immunogenicity Outcomes in People Living With HIV Following Vaccination for COVID-19 (HIV-COV)
Brief Title: Immunogenicity of COVID-19 Vaccination in PLWH
Acronym: HIV-COV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CIHR Canadian HIV Trials Network (Network)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); The Ottawa Hospital (TOH) (Unknown)
Responsible Party: Sponsor
Other Study IDs: CTN 328
Record Dates: First submitted 2021-05-18; First posted 2021-05-20 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PLWH: HIV positive
  Interventions: Biological: COVID-19 Vaccine
- Control: HIV negative
  Interventions: Biological: COVID-19 Vaccine

INTERVENTIONS:
Biological: COVID-19 Vaccine — Any COVID-19 vaccine (1 or more doses)

SUMMARY:
Various facts support the study of COVID-19 vaccine immunogenicity in People Living With HIV (PLWH) at this time: (1) Many PLWH in Canada will be eligible to receive COVID-19 vaccination as they are in a high priority risk group, such as residents or staff of shared living facilities for seniors, health care workers with direct patient contact, aged 70 years of age or older, or adults in Indigenous communities; (2) As vaccines against many other pathogens, it is plausible that the current standard vaccination strategy of COVID-19 is less effective in PLWH; (3) The potential burden of significant COVID-19 infection in PLWH is likely large given many PLWH are aging and have co-morbidities known to predispose to worse COVID-19 outcomes; (4) The vaccine clinical trials which include PLWH63, have stringent exclusion criteria, making results non-generalizable to many PLWH such as those with lower CD4 counts.

With the rapid roll-out of COVID-19 vaccination, many PLWH will be receiving the COVID-19 vaccine. Through vaccination, the provision of the same dosage of antigen stimulation to all individuals will result in a controlled method to measure immune response in PLWH. Therefore, we propose to develop a pan-Canadian cohort of PLWH receiving a COVID-19 vaccine(s) to assess a spectrum of immune responses. We also aim to assess the safety and tolerability of the COVID-19 vaccines in PLWH. These data may provide support for the use of one vaccine product over another and for exploring alternate vaccination strategies in PLWH (i.e., increased dose or double-dose vaccination and so forth).

ELIGIBILITY:
Inclusion Criteria:

* Age >/=16 years (Sites may choose to only enrol adults based on their provincial age of majority)
* HIV positive for HIV group; For HIV negative group, individuals should be immunocompetent and generally in good health (i.e. participants should not have a condition associated with immunodeficiency nor be receiving immunosuppressant medication)
* Receiving at least 1 dose of COVID-19 vaccine, or have received 1 or 2 doses of a COVID-19 vaccine
* Able to provide signed, informed consent
* Able to attend study visits

Exclusion Criteria:

* Signs or symptoms of active COVID-19 infection
* For HIV-uninfected persons: immune-compromising conditions or on medication which suppresses the immune response

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: PLWH and HIV negative controls who have received at least one dose of COVID-19 vaccine
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
immunogenicity of COVID-19 vaccination | 6 months
  as assessed by COVID-19-specific IgG ELISA 6 months following vaccination

SECONDARY OUTCOMES:
Percentage of individuals with COVID-19-specific IgG | 12 months
  Percentage of individuals with COVID-19-specific IgG at 12 months
Percentage of persons whose plasma demonstrate COVID-19 neutralization capacity | 12 months
  as assessed by a pseudotyped viral infection assay
Proportion and activation status of CD4 T cells, CD8 T cells, B cells, natural killer cells and monocytes, pre- and post-vaccination | 12 months
  Proportion and activation status of CD4 T cells, CD8 T cells, B cells, natural killer cells and monocytes, pre- and post-vaccination
Percentage of persons with local or systemic adverse events or use of antipyretic or pain medication within 7 days and 30 days of either first or second injection | 7 and 30 days, post-injection
  Percentage of persons with local or systemic adverse events or use of antipyretic or pain medication within 7 days and 30 days of either first or second injection

OTHER OUTCOMES:
Proportion of individuals with COVID-19-specific IgG at 6 months | 6 months
  stratified by various sub-populations of PLWH
Proportion of individuals with COVID-19-specific IgG at 6 months that cross-recognizes S protein variants of interest, including N501Y and/or E484K. | 12 months
  Proportion of individuals with COVID-19-specific IgG at 6 months that cross-recognizes S protein variants of interest, including N501Y and/or E484K.
Proportion of individuals with COVID-19-specific T cell responses at 6 months, stratified by HLA genotype and immunodominant epitopes in S protein. | 12 months
  Proportion of individuals with COVID-19-specific T cell responses at 6 months, stratified by HLA genotype and immunodominant epitopes in S protein.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Costiniuk, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Curtis Cooper, MD, Principal Investigator — The Ottawa Hospital (TOH); Aslam Anis, PhD, Principal Investigator — CIHR Canadian HIV Trials Network
Locations (3):
- Canada (3):
  - The Ottawa Hospital (TOH), Ottawa, Ontario
  - University Health Network (UHN), Toronto, Ontario
  - Chronic Viral Illness Service (CVIS) McGill University Health Centre (MUHC), Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with Canada's COVID-19 Immunity Task Force (CITF) in accordance with the CITF data sharing agreement. Coded participant data (core data elements: demographics, COVID-19 infection history, health conditions, vaccination, blood testing results) will be deposited into the CITF database every two months for future research concerning COVID-19 and related health outcomes. To request coded centralized data, researchers apply to the CITF Data Access Committee (DAC). The DAC will ask researchers to confirm their intended research activities have received necessary ethics approvals.

REFERENCES:
- [Derived] Costiniuk CT, Singer J, Lee T, Galipeau Y, McCluskie PS, Arnold C, Langlois MA, Needham J, Jenabian MA, Burchell AN, Samji H, Chambers C, Walmsley S, Ostrowski M, Kovacs C, Tan DHS, Harris M, Hull M, Brumme ZL, Lapointe HR, Brockman MA, Margolese S, Mandarino E, Samarani S, Vulesevic B, Lebouche B, Angel JB, Routy JP, Cooper CL, Anis AH; COVAXHIV Study Group. Antibody neutralization capacity after coronavirus disease 2019 vaccination in people with HIV in Canada. AIDS. 2023 Oct 1;37(12):F25-F35. doi: 10.1097/QAD.0000000000003680. Epub 2023 Aug 2. PMID 37534695
- [Derived] Costiniuk CT, Singer J, Lee T, Langlois MA, Arnold C, Galipeau Y, Needham J, Kulic I, Jenabian MA, Burchell AN, Shamji H, Chambers C, Walmsley S, Ostrowski M, Kovacs C, Tan DHS, Harris M, Hull M, Brumme ZL, Lapointe HR, Brockman MA, Margolese S, Mandarino E, Samarani S, Vulesevic B, Lebouche B, Angel JB, Routy JP, Cooper CL, Anis AH; COVAXHIV Study Group. COVID-19 vaccine immunogenicity in people with HIV. AIDS. 2023 Jan 1;37(1):F1-F10. doi: 10.1097/QAD.0000000000003429. Epub 2022 Nov 18. PMID 36476452
- [Derived] Costiniuk CT, Singer J, Langlois MA, Kulic I, Needham J, Burchell A, Jenabian MA, Walmsley S, Ostrowski M, Kovacs C, Tan D, Harris M, Hull M, Brumme Z, Brockman M, Margolese S, Mandarino E, Angel JB, Routy JP, Anis AH, Cooper C. CTN 328: immunogenicity outcomes in people living with HIV in Canada following vaccination for COVID-19 (HIV-COV): protocol for an observational cohort study. BMJ Open. 2021 Dec 16;11(12):e054208. doi: 10.1136/bmjopen-2021-054208. PMID 34916326